CLINICAL TRIAL: NCT05799716
Title: Treating Donors With Intravenous Immunoglobulin to Reduce Donor-Derived Infections
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CT20230313
Record Dates: First submitted 2023-03-13; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Viremia; Bacteremia; Acute Rejection of Renal Transplant
Keywords: IVIG Infection
MeSH Terms: conditions — Viremia; Bacteremia | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IVIG (Experimental)
  Interventions: Drug: IVIG
- Sham (No Intervention)

INTERVENTIONS:
Drug: IVIG — 0.5g/Kg
  Arms: IVIG

SUMMARY:
The goal of this clinical trial is to learn about the benefit of IVIG in donor-derived infections and the potential immunomodulatory effect on transplanted organs. The main questions it aims to answer are:

1. How effective IVIG is in preventing donor-derived infections
2. Does IVIG has potential immunomodulatory effect on transplanted organs

DETAILED DESCRIPTION:
Donor-derived infections are defined as any infection present in the donor that is transmitted to one or more recipient. Donor-derived infections can be categorized into two groups: "expected" and "unexpected" infections. Expected transmissions occur when the donor is known to have an infection, as demonstrated by positive serology or nucleic acid test (NAT) result for cytomegalovirus (CMV), Epstein-Barr virus (EBV) or hepatitis B and C, or positive cultures in the donor at the time of donation. Unexpected transmissions may occur despite current screening strategies and are not expected in the donor at the time of organ placement.

Intravenous immunoglobulins (IVIG) are produced by pooling together of serum immunoglobulins from multiple donors, and are known to have powerful immunomodulatory and anti-inflammatory functions in vitro and in vivo. The goal of this study is to figure out the benefit of IVIG in donor-derived infections and the potential immunomodulatory effect on transplanted organs.

ELIGIBILITY:
Inclusion Criteria:

* Any person approved as a transplant donor with recipient who has never undergone a previous transplantation
* Transplant donor must be 6 years old or older
* They must have provided signed informed consent
* The donors must be willing to contribute samples of blood

Exclusion Criteria:

* Any potential transplant donor who is receiving or have received anti-herpes medication in the past week
* Any potential transplant donor to a recipient who has received a previous solid organ transplant
* Any potential transplant donor who is immunosuppressed due to medical disease and/or immunosuppressive or immunomodulating medications
* Any potential transplant donor who is on corticosteroids

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Next-Generation Sequencing (NGS) Results of Bacteremia or Viremia in Transplant Recipient | 14 days
  NGS is a technology for determining the sequence of DNA or RNA to study genetic variation associated with diseases like bacteremia and viremia.
Incidence of Bacteremia or Viremia in Transplant Recipient | 14 days

SECONDARY OUTCOMES:
Incidence of Acute Rejection in Transplant Recipient | 1 month

IPD SHARING:
Plan to Share IPD: No